CLINICAL TRIAL: NCT03688815
Title: Relationship Between the L-arginine Pathway Metabolites and Dipyridamole Stress Induced Transient Myocardial Ischaemia
Brief Title: Dipyridamole Induced Ischemia and Biomarkers
Status: Completed | Type: Observational
Sponsor: University of Pecs (Other)
Responsible Party: Principal Investigator, Tihamér Molnár, Associate professor, University of Pecs
Other Study IDs: PTE3950
Record Dates: First submitted 2018-09-25; First posted 2018-09-28 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Ischemic Heart Disease; Ischemic Attack
MeSH Terms: conditions — Myocardial Ischemia | interventions — Myocardial Perfusion Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with ischemic heart disease: Patients with ischemic heart disease scheduled for myocardial perfusion scintigraphy were enrolled. Biomarkers were analysed form periferal blood. Patients outcome data were followed up to 5 years.
  Interventions: Diagnostic Test: myocardial perfusion scintigraphy

INTERVENTIONS:
Diagnostic Test: myocardial perfusion scintigraphy — Myocardial perfusion scintigraphy as it is described in the international literature.

SUMMARY:
Analysis of certain biomarkers and transient myocardial perfusion deficit revealed by myocardial perfusion scintigraphy.

DETAILED DESCRIPTION:
The prospectively enrolled patients were followed up to 5 years. Adverse major events (MI, stroke, death) suffered during follow-up were retrospectively analysed.

ELIGIBILITY:
Inclusion Criteria: 1. written informed consent. 2. clinical diagnosis of ischemic heart disease (IHD) -

Exclusion Criteria: 1. refused written informed consent. 2. lost data during follow-up

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients with IHD were enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2010-01-01 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
Myocardial perfusion abnormality | 5 year follow-up after MPS
  Myocardial perfusion was quantified based on myocardial perfusion scintigraphy (MPS).

CONTACTS AND LOCATIONS:
Overall Officials: Tihamer Molnar, MD, Principal Investigator — University of Pecs
Locations (1):
- University of Pecs, Pécs, Baranya, Hungary

IPD SHARING:
Plan to Share IPD: No
IPD sharing plan: publication of data in a peer-reviewed journal

REFERENCES:
- [Derived] Molnar T, Horvath A, Szabo Z, Vamos Z, Doczi T, Illes Z. Detection of silent cerebral microcirculatory abnormalities in patients with manifest ischemic coronary disease: a perfusion brain MRI study combined with dipyridamole stress. Scand Cardiovasc J. 2021 Apr;55(2):97-101. doi: 10.1080/14017431.2020.1821911. Epub 2020 Sep 18. PMID 32945202
- See also: Regulation of Coronary Blood Flow in Health and Ischemic Heart Disease — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC5856234/